CLINICAL TRIAL: NCT05190068
Title: A Multicenter, Open-label, Phase I Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of HMPL-760 in Patients With Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Brief Title: HMPL-760 in Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hutchmed (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2021-760-00CH1
Record Dates: First submitted 2021-12-10; First posted 2022-01-13 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: B-Cell Non-Hodgkin's Lymphoma
Keywords: B-Cell Non-Hodgkin's Lymphoma; Bruton's tyrosine kinase inhibitor
MeSH Terms: conditions — Lymphoma, B-Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Relapsed/refractory B-NHL (Experimental): The starting dose of HMPL-760 is initially set as 50 mg, and then the doses of 100 mg, 200 mg, 300 mg, and 400 mg are escalated successively (this dose gradient is assumed).
  HMPL-760 was administered continuously as a single agent orally every day in sequential 28-day cycles.
  Interventions: Drug: HMPL-760

INTERVENTIONS:
Drug: HMPL-760 — HMPL-760 was administered continuously as a single agent orally every day in sequential 28-day cycles.

SUMMARY:
A Multicenter, Open-label, Phase I Study to Evaluate the Safety, Pharmacokinetics, and Preliminary Efficacy of HMPL-760 in Patients with Relapsed/Refractory B-Cell Non-Hodgkin's Lymphoma

DETAILED DESCRIPTION:
The purpose of this study is to evaluate the safety, tolerability, pharmacokinetics, pharmacodynamics, and preliminary efficacy of HMPL-760 administered orally in subjects with relapsed/refractory B-cell non-Hodgkin lymphoma (B-NHL). Patients with relapsed/refractory B-NHL, including chronic lymphocytic leukemia/small cell lymphoma (CLL/SLL), diffuse large B-cell lymphoma (DLBCL), follicular cell lymphoma (FL), mantle cell lymphoma (MCL), marginal zone lymphoma (MZL), and lymphoplasmacytic/macroglobulinemia (LPL/WM).

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent Form (ICF)
2. Age ≥18 years
3. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1. In the expansion stage, ECOG performance status 0-2
4. Relapsed/refractory patients with histologically confirmed lymphoma

   * CLL confirmed by cytology (flow cytometry)
   * LPL/WM diagnosed by relevant tests including serum, bone marrow, and pathological examinations.
5. Except for CLL and WM, at least one bidimensionally measurable lesion is required by CT scan, which means the largest diameter of lymph node lesions >1.5 cm or extranodal lesions >1.0 cm; For lesions that cannot be well displayed by CT due to anatomical location (such as limb or soft tissue lesions), MRI measurement can be used.
6. Expected survival longer than 24 weeks

Exclusion Criteria:

Patients who met any of the following criteria are excluded from the study:

1. Lymphoma patients with central nervous system (CNS) or leptomeningeal invasion
2. Inadequate organ function of liver and kidney
3. Carcinoma in situ of the breast History of liver disease, including cirrhosis, alcoholism, or currently known active infection with human immunodeficiency virus (HIV), hepatitis B virus (HBV), or hepatitis C virus (HCV)
4. Any anti-tumor therapy including chemotherapy and radiotherapy within 3 weeks prior to the first dose of study drug
5. Within 7 days or approximately 5 half-lives (whichever is longer) prior to the first dose of the investigational drug, received any corticosteroids or approved small molecule targeted anti-cancer therapies.
6. Any monoclonal antibody used for anti-tumor therapy within 4 weeks or 2 half-lives prior to the first dose of study drug, whichever is longer
7. Prior use of any anti-tumor vaccine
8. Prior administration of radioimmunotherapy within 3 months prior to the first dose of study drug
9. Any uncontrolled active infection
10. History of drug-induced interstitial pneumonia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2022-01-04 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
DLTs | Up to 28 days after first dose of study drug.
  Number of subjects with Dose Limiting Toxicities (DLTs) with relapsed/refractory B-cell non-Hodgkin's lymphoma relapsed/refractory B-cell non-Hodgkin's lymphoma
Safety and Tolerability | Baseline up to the end of study
  Number of participants with treatment-related adverse events as assessed by CTCAE v5.0

SECONDARY OUTCOMES:
Objective response rate (ORR) | Baseline up to 6 months after the last patient was enrolled
  Defined as the proportion of patients with CR/Partial response (PR)/CR with incomplete hematologic recovery (CRi)/ partial response with lymphocytosis (PR-L)
Complete response rate (CR rate) | Baseline up to 6 months after the last patient was enrolled
  Defined as the proportion of patients with CR/CRi
Progression-free survival (PFS) | Baseline up to 6 months after the last patient was enrolled
  Defined as the time from the first dose of HMPL-760 to occurrence of Progressive disease (PD) or death, whichever comes first
Time to Response (TTR) | Baseline up to 6 months after the last patient was enrolled
  Defined as the time from the first dose of HMPL-760 to the first objective response
Clinical Benefit Rate (CBR) | Baseline up to 6 months after the last patient was enrolled
  Defined as the proportion of patients with CR/CRi, PR/PR-L and Stable disease (SD)
Duration of Response (DoR) | Baseline up to 6 months after the last patient was enrolled
  Defined as the time from the initial objective response to disease recurrence, progression or death
Overall Survival (OS) | Baseline up to 6 months after the last patient was enrolled
  Defined as the time from the first dose to death due to any cause

CONTACTS AND LOCATIONS:
Overall Officials: Weili Zhao, Ph.D, Principal Investigator — Shanghai Jiao Tong University School of Medicine
Locations (22):
- China (22):
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University, Xiameng, Fujian
  - Sun Yat-sen University Cancer Center, Guangzhou, Guangdong
  - Guangxi Medical University cancer Hospital & Guangxi Cancer Institute, Nanning, Guangxi
  - Affiliated Hospital of Chengde Medical University, Chengde, Hebei
  - Henan Cancer Hospital, Zhengzhou, Henan
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Chenzhou First People's Hospital, Chenzhou, Hunan
  - First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Jiangxi Cancer Hospital, Nanchang, Jiangxi
  - Jilin Cancer Hospital, Changchun, Jilin
  - The Second Affiliated Hospital of Dalian Medical University, Dalian, Liaoning
  - The First Hospital of China Medical University, Shenyang, Liaoning
  - Harbin Medical University Cancer Hospital, Harbin, Longjiang Hei
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Heping Hospital Affiliated to Changzhi Medical College, Changzhi, Shanxi
  - Shanxi Bethune Hospital, Taiyuan, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - Affiliated Hangzhou First People's Hospital ,Zhejiang University School of Medicine, Hangzhou, Zhejiang
  - Chongqing university cancer hospital, Chongqing
  - Ruijin Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai